CLINICAL TRIAL: NCT06969053
Title: Evaluation of Mindfulness Intervention Therapy in Treating Chronic Insomnia (CI) With Comorbid Anxiety
Brief Title: Effect of MIT for CI With Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI+CA-MIT
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chronic Insomnia; Anxiety Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIT + SHE (Experimental)
  Interventions: Behavioral: Mindfulness Intervention Therapy plus Sleep Hygiene Education
- SHE only (Active Comparator)
  Interventions: Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Mindfulness Intervention Therapy plus Sleep Hygiene Education — Participants will receive a 6-week program combining Mindfulness Intervention Therapy (MIT) and Sleep Hygiene Education (SHE). MIT includes body scan, mindful breathing, breathing space exercises, mindful walking, sitting meditation, loving-kindness meditation, and development of a personalized mindfulness practice plan. Sessions are conducted daily for 50 minutes. SHE provides structured guidance on optimizing sleep schedules, bedroom environment, and reducing stimulants such as caffeine and alcohol.
  Arms: MIT + SHE
Behavioral: Sleep Hygiene Education — Participants will receive Sleep Hygiene Education (SHE) alone for 6 weeks. SHE involves education on maintaining consistent sleep schedules, creating a sleep-conducive environment, reducing stimulant use (e.g., caffeine, alcohol), and promoting healthy daily routines to improve sleep quality.
  Arms: SHE only

SUMMARY:
This randomized controlled trial aims to investigate the efficacy of Mindfulness Intervention Therapy (MIT) in treating Chronic Insomnia (CI) comorbid with anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Insomnia Disorder according to DSM-5 criteria.
2. Pittsburgh Sleep Quality Index (PSQI) total score > 5.
3. Age 8 years or older.
4. Educational level of at least junior high school.
5. Voluntarily agree to participate and provide written informed consent.
6. Presence of anxiety symptoms, defined as Hamilton Anxiety Rating Scale (HAMA) score ≥ 14.

Exclusion Criteria:

1. Presence of severe physical illnesses or major psychiatric disorders, or at risk of suicide.
2. Diagnosed or suspected of having sleep breathing disorders, restless legs syndrome, circadian rhythm sleep disorders, or engaged in shift work.
3. Pregnant or breastfeeding women.
4. Currently undergoing any psychological therapy.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
The change of Pittsburgh Sleep Quality Index (PSQI) total scores from baseline to 6 weeks | Baseline, 6 weeks
  The PSQI consists of 7 factors ranging from 0 to 3 points, and the total score ranges from 0 to 21 with higher scores indicating poorer quality.

SECONDARY OUTCOMES:
The change of Insomnia severity index (ISI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The ISI reporting insomnia symptoms severity consists of 7-items on a 5-point Likert scale, and the total score ranges from 0 to 28 with higher scores indicating more severe insomnia.
The change of sleep efficiency from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  Sleep efficiency is assessed with the Carney (2012) consensus sleep diary. This is measured in percentage (higher scores indicating better sleep efficiency).
The change of Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The DBAS assessing sleep related cognitions in 16 items rated on a 10-point Likert scale, and the total score ranges from 0 to 160 with higher scores indicating more intensive dysfunctional beliefs.
The change of Snaith-Hamilton Pleasure Scale (SHAPS) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The SHAPS assessing anhedonia consists of 14 items, and the total score ranges from 14 to 56 with higher scores indicating more serious the anhedonia.
The change of Short Form 36 (SF-36) total scores from baseline to 6 weeks, 3 months, 6 months, 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months.
  The SF-36 quantifying the quality of life in relation to health status consists of 36-items with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The total score ranges from 0-100 (the worst possible to the most possible).
The change of Patient Health Questionnaire-4 (PHQ-4) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-4 comprises a 2-item depression scale and a 2-item anxiety scale. Each instrument can reach values from 0-6. Higher Scores are indicating higher distress.
The change of Beck Depression Inventory (BDI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BDI assessing the existence and severity of symptoms of depression consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe depressive symptoms.
The change of Beck Anxiety Inventory (BAI) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The BAI assessing the existence and severity of symptoms of anxiety consists of 21 items, and the total score ranges from 0 to 63 with higher scores indicating more severe anxiety.
The change of Patient Health Questionnaire-15 (PHQ-15) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PHQ-15 measuring somatic distress consists of 15 items, and the total score ranges from 0 to 30 with higher scores indicating more severe somatic distress.
The change of 5-item Perceived Deficits Questionnaire-Depression (PDQ-D-5) total scores from baseline to 6 weeks, 3 months, 6 months, and 12 months | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The PDQ-D-5 assessing perceived cognitive deficits from the patient's perspective consists of 5 items, and the total score ranges from 0 to 20 with higher scores indicating greater perceived deficit.
The change of Life Events Scale (LES) total scores from baseline to 3 months, 6 months, 12 months, 18 months, and 24 months. | Baseline, 6 weeks, 3 months, 6 months, and 12 months
  The LES assessing the perceived stress and number of stressful life events experienced consists of 48 items which are classified into three dimensions: family life events (28 items), work and study events (13 items), and social events (7 items) with higher scores in LES perceived greater stressfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028